CLINICAL TRIAL: NCT02486666
Title: A Pilot Feasibility And Safety Multicenter Trial Of Administering Weight Adjusted Fixed Dose Of Low Molecular Weight Heparin (Enoxaparin) To Neonates and Children With Thrombosis (FiXET)
Brief Title: Pilot Feasibility and Safety of Administering Weight Adjusted Fixed LMWH Dose
Acronym: FiXET
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: IWK Health Centre (Other); Children's Hospital of Philadelphia (Other); Children's Hospital of Eastern Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HamiltonHSC
Record Dates: First submitted 2015-05-14; First posted 2015-07-01 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Venous Thromboembolism
Keywords: Enoxaparin; thrombosis; neonate; children; RCT
MeSH Terms: conditions — Venous Thromboembolism; Thrombosis | interventions — Enoxaparin; enoxaparin sodium

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm (Experimental): Experimental Arm:patients will not have any dose titration regardless of anti-Xa level.
  Premature neonates will receive enoxaparin 2.0 mg/kg/dose rounded to nearest whole mg twice daily, while term neonates will receive enoxaparin 1.7 mg/kg/dose rounded to nearest whole mg twice daily. Children≥1 month corrected age will receive 1.5 mg/kg/dose twice daily (maybe rounded +/- 10% for convenience of dosing) while children≥2 month corrected age will receive 1.0 mg/kg/dose twice daily (maybe rounded +/- 10% for convenience of dosing).
  Interventions: Drug: Enoxaparin
- Control Arm (Other): Control Arm: patients who will have dose titration based on anti-Xa levels to maintain a therapeutic range of 0.5-1.0 u/mL (standard of care).
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — WEIGHT ADJUSTED FiXED DOSE OF LOW MOLECULAR WEIGHT HEPARIN (ENOXAPARIN) TO NEONATES AND CHILDREN WITH THROMBOSIS (FiXET)
  Other Names: Enoxaparin sodium

SUMMARY:
Background Enoxaparin is a commonly used low molecular weight heparin (LMWH) for the treatment of neonatal and children thrombosis that is monitored with anti-factor Xa (anti-Xa) levels. However, this therapeutic range of anti-Xa (0.5 - 1.0 u/ml) was extrapolated from adult studies. The burden of pain to neonates due to venipunctures and of resources to the health care system also warrants an evidence-based review to assess the utility of monitoring LMWH therapy with anti-Xa levels.

Methods/Design This is a prospective pilot, feasibility and safety multicenter, randomized controlled trial to compare the approach of treating thrombosis in neonates and children with enoxaparin using weight adjusted fixed dose to variable dose titrated to maintain a pre-determined anti-Xa range (0.5-1.0 u/mL). We plan to recruit 20 neonates and children over the study period, who will be randomized within their first week of anti-coagulation treatment. Key feasibility outcomes include screening/recruitment ratio, monthly recruitment rate, and completeness of data collection. We will also measure the safety outcome of bleeding as well as comment on efficacy of resolution of thrombosis as a secondary outcome.

Discussion The administration of weight adjusted fixed dose of enoxaparin without anti-Xa monitoring has the potential to reduce pain from multiple venipunctures in neonates and children as well as resources used in their already complex care. The results of the FiXET trial will set the framework for a larger multicenter randomized controlled trial to compare the efficacy of administering enoxaparin to neonates and children without monitoring to the current conventional approach of routine monitoring with anti-Xa levels.

DETAILED DESCRIPTION:
1. Scientific Rationale Enoxaparin is a commonly used low molecular weight heparin (LMWH) for the treatment of neonatal and children thrombosis that is monitored with anti-factor Xa (anti-Xa) levels. However, this therapeutic range of anti-Xa (0.5 - 1.0 u/ml) was extrapolated from adult studies. The burden of pain to neonates and children due to venipunctures and of resources to the health care system also warrants an evidence-based review to assess the utility of monitoring LMWH therapy with anti-Xa levels. This FiXET trial is to compare the approach of treating thrombosis in neonates and children with enoxaparin using weight adjusted fixed dose to variable dose titrated to maintain a pre-determined anti-Xa range (0.5-1.0 u/mL). We plan to recruit 20 neonates and children over the study period, who will be randomized within their first week of anti-coagulation treatment. Key feasibility outcomes include screening/recruitment ratio, monthly recruitment rate, and completeness of data collection. We will also measure the safety outcome of bleeding as well as comment on efficacy of resolution of thrombosis as a secondary outcome.

   1.1 Potential Risk and Benefits The administration of weight adjusted fixed dose of enoxaparin without anti-Xa monitoring has the potential to reduce pain from multiple venipunctures in neonates and children as well as resources used in their care. The results of the FiXET trial will provide preliminary clinical data regarding the feasibility and safety of this approach to anticoagulation treatment in neonates and children. It will also provide a preliminary idea about the efficacy of such an approach. This trial, if successful, will set groundwork for a larger multicenter randomized controlled trial to compare the efficacy of administering enoxaparin to neonates and children without monitoring to the current conventional approach of routine monitoring with anti-Xa levels.
2. Study Objectives The aim of this trial is to determine the feasibility and safety of doing a randomized control trial to compare the approach of treating thrombosis in neonates and children with enoxaparin using weight adjusted fixed dose to variable dose titrated to maintain a pre-determined anti-Xa range (0.5-1.0 u/mL).
3. Eligibility Criteria Four or more tertiary hospitals will participate in this trial. We plan to recruit a total of 20 patients based on the following protocol-defined inclusion and exclusion criteria.
4. Study Design FiXET trial is a prospective pilot, feasibility and safety multicenter, randomized controlled trial. Recruitment will start following institutional REB approval. This will occur over 1year per centre and may take up to 2 years. Analysis and dissemination will occur after this period of time.

   4.1 Study Endpoints

   Primary Objective The primary outcome of this trial is to assess feasibility and safety, as defined below, of administering a weight adjusted fixed dose of enoxaparin to neonates and children with thrombosis.

   Feasibility criteria
   * At least 5 subjects can be recruited in each participating centre over the study period
   * At least 50% of all approached patients can be recruited
   * Complete data collection and follow-up of at least 90% of all recruited subjects

   Safety criteria

   - No more than 20% of subjects are removed from the study due to 1) low or high anti-Xa levels, or 2) major bleeding

   Major bleeding will be defined as (i) fatal bleeding; (ii) clinically overt bleeding resulting associated with a decrease in hemoglobin of 20 g/L (2 g/dL) in a 24 hour period; (iii) bleeding into a critical organ (intracranial, pulmonary or retroperitoneal); or bleeding requiring surgical intervention [17].

   Minor bleeding will be defined as any overt or macroscopic evidence of bleeding that does not fulfill criteria for major bleeding [17].

   Secondary Objective Secondary outcome measures include 1) efficacy in resolution of thrombosis; 2) mean anti-Xa levels; 3) number of enoxaparin dose adjustments required in the control arm; and 4) number of venipuncture attempts for blood sampling in patients.
5. Expected Duration of Participant Participation The duration of enoxaparin therapy will be 6 weeks to 6 months at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria

* Birth to under 18 years of age at the diagnosis of thrombosis event
* Diagnosis of deep vein thrombosis confirmed by either venography or ultrasound, pulmonary embolism confirmed by ventilation perfusion scan or spiral CT scan or pulmonary angiogram, clinically stable cerebral sinovenous thrombosis confirmed with magnetic resonance imaging, or cardiac thrombosis diagnosed by echocardiogram.
* The treating team has decided to initiate anti-coagulation therapy

Exclusion Criteria

* Platelet count < 50x109/L;
* Hemorrhage or high risk of bleeding with the use of anticoagulation therapy;
* Creatinine > 1.5x upper limit of normal;
* Liver dysfunction associated with coagulopathy leading to a clinically relevant bleeding risk;
* Documented history of heparin induced thrombocytopenia;
* Known contraindication to heparin

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-03; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruiting at least 5 subjects over the study period per center | 12 - 24 months
  * Number of Participants from each participating center
  * Rate of recruitment per approaching
  * Rate of completed data collection and follow-up per all recruited subjects These variables will be combined to reflect the feasibility of trial recruitment
Safety of administering a weight adjusted fixed dose of enoxaparin to neonates and children with thrombosis | 12 - 24months
  - Percentage of subjects removed from the study due to 1) low or high anti Xa levels or 2) major bleeding

SECONDARY OUTCOMES:
Efficacy in resolution of thrombosis | 12-24 months
  -Rate of thrombosis resolution
Safety of anticoagulation | 12-24 months
  * Mean anti-Xa levels
  * Number of Enoxaparin dose adjustments in the control arm
  * Number of venipuncture attempts for blood sampling These Categorical variables will be combined to analyze the safety of this FiXET dose anticoagulation therapy on patients

CONTACTS AND LOCATIONS:
Overall Officials: Mihir Bhatt, MD, Principal Investigator — HHSC/McMaster Children's Hospital
Locations (4):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States
- Canada (3):
  - IWK Health Center, Halifax, Nova Scotia
  - HHSC/McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No